CLINICAL TRIAL: NCT04927806
Title: The Effectiveness of Antimicrobial Breathing System on the Presence of Multidrug-resistant Organisms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fu Jen Catholic University (Other)
Responsible Party: Principal Investigator, Ke-Yun, Chao, Group leader of Respiratory Therapists, Fu Jen Catholic University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: PL-202108037M
Record Dates: First submitted 2021-06-09; First posted 2021-06-16 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Bacterial Contamination
Keywords: Bacterial contamination; nosocomail infection; bacterial detection rate

STUDY DESIGN:
Intervention Model Description: In this study, we conduct a cluster-randomized crossover, multicenter trial.There are two groups:
  1. Control group: standard ventilator circuit in odd number month.
  2. Experimental group: Silver Knight in even number month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SilverKnight group (Experimental): Silver Knight is an anti-microbial additive that uses silver ions to disrupt the normal enzymatic activities of bacteria
  Interventions: Device: Silver Knight
- Control group (No Intervention): The control group uses standard ventilator circuits.

INTERVENTIONS:
Device: Silver Knight — Silver Knight breathing systems are all validated for up to seven days use, and remain active, in unopened packaging, for up to five years. Silver Knight is proven to help reduce the incidence of MRSA infection and other organisms including:
  * Staphyloccus epidermis
  * Pseudomonas aeruginosa
  * Klebsiella pneumoniae
  * Acinetobacter calcoaceticus
  * Escherichia coli
  Arms: SilverKnight group

SUMMARY:
The aim of this study is to investigates the effectiveness of antimicrobial breathing system on multidrug-resistant organisms (MDRO).

DETAILED DESCRIPTION:
Background:

Cross transmission via skin contact and environmental media is the main route for common outbreak of health care-associated infection which more likely to be improved or prevented by infection control program. Silver Knight uses silver ions to disrupt the normal enzymatic activities of bacteria for reducing microbial growth within, and on, the surface of the breathing systems. It functions as a safe, quick and effective catalyst to deactivate pathogenic bacteria and prevent their proliferation. However, there was no study comparing the standard ventilator circuit with Silver Knight. This study focuses on the effectiveness of antimicrobial breathing system in MDRO which including carbapenem-resistant, vancomycin-resistant and multi-drug resistant.

Study Design:

This is a prospective, randomized study in a single hospital in the intensive care unit.

Methods:

In this study, we conduct a cluster-randomized crossover, single-centre trial. There are two groups:

1. Control group: standard ventilator circuit in odd number month.
2. Experimental group: Silver Knight in even number month This study is expected to recruit 200 subjects. During this period, the ventilator circuits are all routinely used, only the tubing will not be discarded after use for specimen collection.And the MDRO on the surfaces of ventilator circuits will be analyzed and evaluated.

Effect:

We expect the antimicrobial breathing system could be more effectively than the standard ventilator circuit. The policy related to current ventilator circuit will be revised according to the results of this study.

Key words:

Antimicrobial Breathing system, ventilator circuits, multidrug-resistant organisms (MDRO)

ELIGIBILITY:
Inclusion Criteria:

* mechanical ventilators in Medisive CareUnit (MICU)

Exclusion Criteria:

* Using ventilators for less than seven days

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
bacterial contamination | one month
  comparison of the two ventilator systems

SECONDARY OUTCOMES:
bacterial detection rate | one month
  comparison of the two ventilator systems

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Lun Liu, MD, Principal Investigator — Department of Emergency and Critical Care Medicine, Fu Jen Catholic University Hospital
Locations (1):
- Fu Jen Catholic University Hospital, Fu Jen Catholic University, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zilahi G, Artigas A, Martin-Loeches I. What's new in multidrug-resistant pathogens in the ICU? Ann Intensive Care. 2016 Dec;6(1):96. doi: 10.1186/s13613-016-0199-4. Epub 2016 Oct 6. PMID 27714706
- [Derived] Chao KY, Liu WL, Chen CY, Su CH, Yang SH, Huang YT. Bacterial Colonization of Silver-Additive Ventilator Circuit in Patients Receiving Mechanical Ventilation: A Randomized Controlled Trial. Clin Respir J. 2025 Mar;19(3):e70058. doi: 10.1111/crj.70058. PMID 40052538